CLINICAL TRIAL: NCT02541578
Title: Physiological Complexity of Gait Over the First Six Months Post Stroke
Status: Completed | Type: Observational
Sponsor: University of Indianapolis (Other)
Collaborators: Seattle University (Unknown)
Responsible Party: Principal Investigator, Stephanie Miller, Professor, University of Indianapolis
Other Study IDs: 0721
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Stroke, Acute
Keywords: stroke, acute; gait, complexity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Physiological complexity of gait, a measure of the interaction of multiple control mechanisms for walking within a biological system, is decreased in persons with chronic stroke compared to those without disability. Thus, it is assumed that the quantification of gait complexity represents the adaptability and health of the individual. However, it is unknown if the level of gait-related complexity improves over time with recovery from stroke. Therefore, the primary purpose of this study is to determine if the physiological complexity of gait changes over the first six months post stroke within the contemporary healthcare environment. Secondary aims include 1) determining if there is a difference between the amount of physiological complexity of gait and lateralization of hemispheric damage after stroke and 2) exploring the relationship of complexity to lower extremity motor impairment, walking speed and balance. Sixty individuals within one month post stroke from the greater Indianapolis area will be recruited for this prospective, longitudinal outcomes study. Testing sessions will occur at intervals across the first six months post stroke: within 1 month, at 3 months, and at 6 months post stroke. During each testing session, participants will complete a 2-minute walking task during which accelerometer signals from wireless inertial measurement units will be collected and converted to sample entropy to quantify the physiological complexity of gait. Additionally, measures to quantify lower extremity motor impairment, walking speed and balance will be collected and analyzed. Changes in complexity of gait from early to later stages of stroke recovery may serve as a foundation for prognosticating outcomes, such as predicting capacity for community mobility and/or risk of fall. The proposed study will meet a critical need to develop methods that differentiate among capacities for adapting movement patterns in individuals with neurological dysfunction. This work will ultimately build upon evidence that will assist therapists in tailoring interventions in such a way to optimize function.

ELIGIBILITY:
Inclusion Criteria:

* within 1-month post unilateral, cortical, ischemic stroke
* has only experienced one stroke
* between the ages of 21-80
* able to walk a short distance (at least 14 meters) on level surfaces without physical assistance, with or without the use of an assistive device and/or orthosis
* able to follow at least two-step verbal instructions
* available for the entire period of the study (5-6 months)

Exclusion Criteria:

* hemorrhagic stroke
* bilateral hemispheric stroke
* stroke in the brainstem or cerebellum
* pre-existing neurological or current musculoskeletal conditions that would limit gait ability separate from the effects of stroke
* complications from other health conditions that could influence walking

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 60 adults with acute stroke will be enrolled in this prospective, longitudinal cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in physiological complexity index of gait over 6 months | Within 1 month, 3 months and 6 months post stroke
  Participants will complete a 2-minute walking task on a level indoor surface using their preferred pace during which accelerometer signals from wireless inertial measurement units will be collected. This data will be used to calculate multivariate multiscale sample entropy in order to quantify the complexity index in all lower segments (thigh, shank, foot) and pelvis during gait.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Miller, PT, PhD, NCS, Principal Investigator — University of Indianapolis
Locations (1):
- University of Indianapolis, Krannert School of Physical Therapy, Indianapolis, Indiana, United States